CLINICAL TRIAL: NCT00334672
Title: Hemophagocytic Lymphohistiocytosis
Brief Title: Combination Chemotherapy Followed By Donor Stem Cell Transplant in Treating Patients With Hemophagocytic Lymphohistiocytosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Children's Cancer and Leukaemia Group (Other)
Organization: National Cancer Institute (NCI) (NIH)
Masking: None | Purpose: Treatment
Other Study IDs: CDR0000481605; CCLG-LCH-2006-02; EU-20619; UKCCSG-HLH-2004; EUDRACT-2005-002187-28
Record Dates: First submitted 2006-06-07; First posted 2006-06-08 (Estimated); Last update posted 2013-09-17 (Estimated); Status verified 2009-06

CONDITIONS: Nonneoplastic Condition
Keywords: hemophagocytic lymphohistiocytosis
MeSH Terms: conditions — Lymphohistiocytosis, Hemophagocytic | interventions — Antilymphocyte Serum; Busulfan; Cyclophosphamide; Cyclosporine; Dexamethasone; Etoposide; Methotrexate; Mycophenolic Acid; Hydrocortisone; Biopsy

INTERVENTIONS:
Biological: anti-thymocyte globulin
Drug: busulfan
Drug: cyclophosphamide
Drug: cyclosporine
Drug: dexamethasone
Drug: etoposide
Drug: methotrexate
Drug: mycophenolate mofetil
Drug: therapeutic hydrocortisone
Other: laboratory biomarker analysis
Procedure: allogeneic hematopoietic stem cell transplantation
Procedure: biopsy

SUMMARY:
RATIONALE: Drugs used in chemotherapy work in different ways to stop the growth of hemophagocytic lymphohistiocytosis cells, either by killing the cells or by stopping them from dividing. Giving more than one drug (combination chemotherapy) may kill more hemophagocytic lymphohistiocytosis cells. A donor stem cell transplant may be able to replace blood-forming cells that were destroyed by chemotherapy. Sometimes the transplanted cells from a donor can make an immune response against the body's normal cells. Cyclosporine and methotrexate may stop this from happening.

PURPOSE: This phase III trial is studying how well combination chemotherapy followed by a donor stem cell transplant works in treating patients with hemophagocytic lymphohistiocytosis.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Provide and evaluate revised induction and maintenance therapy comprising etoposide, dexamethasone, and cyclosporine, in terms of achieving and maintaining an acceptable clinical condition in order to perform a curative allogeneic hematopoietic stem cell transplantation (AHSCT), in patients with primary inherited or severe and persistent secondary hemophagocytic lymphohistiocytosis (HLH).
* Evaluate and improve the outcome of AHSCT with various types of donors.
* Determine the prognostic importance of the state of remission at the time of AHSCT.
* Evaluate the neurological complications, in terms of early neurological alterations and cerebrospinal fluid (CSF) findings, in patients treated with this regimen.

Secondary

* Improve the understanding of the pathophysiology of HLH by conducting biological studies of genetics and cytotoxicity in these patients, including genotype-phenotype studies and the prognostic value of natural killer (NK) cell activity subtyping.

OUTLINE: This is a multicenter study.

* Induction therapy (weeks 1-8): Patients receive etoposide IV over 1-3 hours twice weekly in weeks 1 and 2 and then once weekly in weeks 3-8. Patients also receive dexamethasone IV or orally once daily and cyclosporine IV or orally twice daily in weeks 1-8. Patients with clinically evident, progressive neurological symptoms or an abnormal cerebrospinal fluid (CSF) (cell count and protein) that has not improved after 2 weeks of induction therapy undergo intrathecal therapy comprising methotrexate and hydrocortisone once weekly in weeks 3-6.

Patients are evaluated after 8 weeks of induction therapy. Patients with primary (i.e., familial) hemophagocytic lymphohistiocytosis (HLH) or genetic evidence of HLH proceed to maintenance therapy. Patients with severe and persistent secondary (i.e., nonfamilial) HLH and no genetic evidence of HLH proceed to maintenance therapy only if their disease is still active after induction therapy. Patients with nonfamilial HLH and no genetic evidence of HLH who have achieved complete remission (CR) discontinue treatment. If their disease reactivates, they may then proceed to allogeneic hematopoietic stem cell transplantation (AHSCT).

* Maintenance therapy (weeks 9-40): Patients receive dexamethasone IV on days 1-3 in weeks 10, 12, 14, 16, 18, 20, 22, 24, 26, 28, 30, 32, 34, 36, 38, and 40; etoposide IV over 1-3 hours once in weeks 9, 11, 13, 15, 17, 19, 21, 23, 25, 27, 29, 31, 33, 35, 37, and 39; and cyclosporine IV or orally twice daily in weeks 9-40.

After completion of maintenance therapy, patients with primary (i.e., familial) HLH, severe and persistent secondary (i.e., nonfamilial) HLH, or reactivating disease proceed to AHSCT. Patients with nonfamilial HLH who have completed maintenance therapy, but do not go on to receive AHSCT, may be recommended for additional maintenance therapy at the discretion of the treating physician.

* AHSCT:

  * Preparative regimen: Patients receive a preparative regimen comprising busulfan orally or IV four times daily on days -8 to -5, etoposide IV over 6 hours on day -4, and cyclophosphamide IV over 1 hour on days -3 and -2. Patients who are undergoing unrelated AHSCT, also receive antithymocyte globulin (ATG) IV over 12 hours on days -3 to -1.
  * Transplantation: Patients undergo AHSCT on day 0.
  * Graft-versus-host disease prophylaxis: Beginning on day -1, patients receive cyclosporine IV continuously and then orally, when tolerated, once daily for 6-12 months. Patients also receive methotrexate* IV on days 1, 3, and 6.

NOTE: *As a substitute for methotrexate, patients may receive oral mycophenolate mofetil twice daily on days 0-40, followed by a taper and discontinuation.

Patients undergo periodic blood collection and bone marrow biopsies for biological studies.

After completion of study treatment, patients are followed periodically for up to 5 years.

PROJECTED ACCRUAL: A total of 288 patients will be accrued for this study.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Newly diagnosed hemophagocytic lymphohistiocytosis (HLH) meeting 1 of the following criteria*:

  * Diagnosis by molecular/genetic methods
  * Diagnosis by meeting 5 out of 8 of the following criteria:

    * Clinical criteria:

      * Fever
      * Splenomegaly
    * Laboratory criteria:

      * Cytopenias affecting ≥ 2 of 3 lineages in the peripheral blood, including the following:

        * Hemoglobin < 9.0 g/dL (< 10.0 g/dL in infants < 4 weeks of age)
        * Platelet count < 100,000/mm^3
        * Neutrophil count < 1,000/mm^3
      * Hypertriglyceridemia and/or hypofibrinogenemia:

        * Fasting triglycerides ≥ 3.0 mmol/L (i.e., ≥ 265 mg/dL)
        * Fibrinogen ≤ 1.5 g/L
    * Histopathologic criteria:

      * Hemophagocytosis in bone marrow, spleen, or lymph nodes

        * No evidence of malignancy
    * New diagnostic criteria:

      * Low or absent natural killer (NK) cell activity
      * Ferritin ≥ 500 mcg/L
      * Soluble CD25 (i.e., soluble interleukin-2 receptor) ≥ 2,400 U/mL NOTE: *Patients who do not meet the diagnostic criteria for HLH but who have a strong clinical suspicion of HLH may be eligible at the discretion of the investigator
* Primary HLH (i.e., familial hemophagocytic lymphohistiocytosis [FLH]) OR secondary HLH (i.e., severe acquired form of HLH)
* Acceptable donor meeting 1 of the following criteria:

  * HLA-identical related donor
  * Matched unrelated donor
  * Mismatched unrelated donor
  * Familial haploidentical donor

PATIENT CHARACTERISTICS:

* Not specified

PRIOR CONCURRENT THERAPY:

* No prior cytotoxic treatment for HLH
* No prior cyclosporine treatment for HLH

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 288 (Estimated)
Dates: Start 2006-03; Primary Completion 2010-11 (Estimated)

PRIMARY OUTCOMES:
Survival

CONTACTS AND LOCATIONS:
Overall Officials: Vasanta Nanduri, MD, Study Chair — Watford General Hospital
Locations (13):
- United Kingdom (13):
  - Birmingham Children's Hospital, Birmingham, England
  - Institute of Child Health at University of Bristol, Bristol, England
  - Addenbrooke's Hospital, Cambridge, England
  - Watford General Hospital, Herts, England
  - Leeds Cancer Centre at St. James's University Hospital, Leeds, England
  - Royal Liverpool Children's Hospital, Alder Hey, Liverpool, England
  - Great Ormond Street Hospital for Children, London, England
  - Royal Manchester Children's Hospital, Manchester, England
  - Children's Hospital - Sheffield, Sheffield, England
  - Southampton General Hospital, Southampton, England
  - Royal Aberdeen Children's Hospital, Aberdeen, Scotland
  - Royal Hospital for Sick Children, Edinburgh, Scotland
  - Royal Hospital for Sick Children, Glasgow, Scotland